CLINICAL TRIAL: NCT05255341
Title: Clinical and Radiographic Evaluation of the Effect of Socket Preservation Using the Roll Pedicle Connective Tissue Graft With Bovine Bone: A Case Series Trial.
Brief Title: Clinical and Radiographic of the Effect of Socket Preservation Using the Roll Pedicle Connective Tissue Graft With Bovine Bone: A Case Series Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Magdy Salem Amen Eladly, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: roll pedicle graft
Record Dates: First submitted 2022-02-08; First posted 2022-02-24 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-02

CONDITIONS: Socket Preservation
Keywords: socket preservation; vascularized interpositional connective tissue graft; alveolar ridge preservation techniques; bovine bone graft; roll pedicle graft

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- roll pedicle connective tissue graft with bovine bone (Experimental): 1. sulcular incisions were performed on the buccal and lingual aspects of the teeth to be extracted
  2. Atraumatic extraction was made by periotome.
  3. After tooth extraction the soft tissue was reflected at least 4 mm beyond the alveolar crest margin and the socket was filled with bovine derived xenograft and covered with roll pedicle connective tissue graft as a barrier membrane.
  4. This pedicle is rolled under the buccal mucosa.The palatal connective tissue pedicle graft was outlined by full thickness incision along the oblique incision line, and parallel incision given from the mesial line angle of target place and reflected coronally up to the crest of the ridge defect. then a partial thickness incision was made extending beyond the line angles of adjacent incisors and mucogingival junction, leaving the periosteum on the bone.
  5. the pedicle graft was rolled from the apical end and secured with interrupted sutures to the labial flap.
  Interventions: Procedure: roll pedicle connective tissue graft with bovine bone

INTERVENTIONS:
Procedure: roll pedicle connective tissue graft with bovine bone — rotated pedicle connective tissue graft together with bovine bone applied for socket preservation after tooth extraction
  Other Names: vascularized interpositional connective tissue graft

SUMMARY:
After tooth extraction, the residual alveolar ridge generally provides limited bone volume because of ongoing, progressive bone resorption. Healing events within post-extraction sockets reduce the dimensions of the socket over time. Therefore, socket preservation became an indispensable procedure as well as fundamental to prevent bone loss following tooth extraction. Preservation, by the name, is the maintenance of the socket, which is essentially the height and width of the gap that is left after the tooth is removed. It is done by placing a graft material or scaffold immediately into the socket of an extracted tooth to presto preserve bone height, width and density

DETAILED DESCRIPTION:
Investigator evaluate the clinical and radio graphic effect of roll pedicle connective tissue graft as a barrier membrane together with bovine bone in alveolar ridge preservation in extraction sockets.

ELIGIBILITY:
Inclusion Criteria:

* • patients with healthy systemic condition.

  * Adult patients ˃ 18 years old.
  * hopeless teeth that need tooth or root extraction in the maxillary esthetic zone.
  * Alveolar socket Grade I and II.
  * Normal platelet counts according to complete blood count (CBC) test done in the screening stage.

Exclusion Criteria:

* Acute infection at the extraction site

  * Smokers ˃ 10 cigarettes / day.
  * Medications that may interfere with wound healing
  * History of treatment with bisphosphonates.
  * History of allergic reaction

Ages: 27 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-09-16 (Actual)

PRIMARY OUTCOMES:
width of alveolar bone | changes in the Width of alveolar bone were measured at 3& 5 mm at baseline,3 months and 6 months
  Two holes will be made in the acrylic stent (3mm and 5 mm below the alveolar crest) on the buccal and palatal extensions within the midline of the tooth to be extracted.
  The buccopalatal width of the alveolar ridge will be measured at the two assigned points using bone caliper at baseline and 6 months post extraction

SECONDARY OUTCOMES:
gingival thickness | changes in the gingival thickness were measured at 3 & 5mm at (baseline,3 months and 6 months)
  Two holes will be made in the acrylic stent (3mm and 5 mm below the alveolar crest) on the buccal and palatal extensions within the midline of the tooth to be extracted.
  The gingival thickness will be evaluated by William's graduated periodontal probe inserted horizontally perpendicular to the alveolar bone at the two assigned holes labially/buccally at baseline and 6 Two holes will be made in the acrylic stent (3mm and 5 mm below the alveolar crest) on the buccal and palatal extensions within the midline of the tooth to be extracted.
  The gingival thickness will be evaluated by William's graduated periodontal probe inserted horizontally perpendicular to the alveolar bone at the two assigned holes labially/buccally at baseline and 6 months post extraction.
  months post extraction.
height of the alveolar crest | changes in height of alveolar crest were measured at baseline, 3 months and 6 months
  Crestal bone height was measured to determine the amount of bone at gain using digora soft ware

CONTACTS AND LOCATIONS:
Overall Officials: noha magdy salem amin, Principal Investigator — cairo university- faculty of dentistry
Locations (1):
- Faculty of Dentistry -Cairo University, Giza, Egypt